CLINICAL TRIAL: NCT01409369
Title: A Single-Center, Open-Label, Two-Period Crossover Study to Investigate the Effect of Multiple Doses of Activated Charcoal on the Pharmacokinetics of a Single Oral Dose of RO4995819 in Healthy Subjects.
Brief Title: A Study on The Effect of Multiple Doses of Activated Charcoal on The Pharmacokinetics of a Single Dose of RO4995819
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None
Other Study IDs: BP25485; 2011-000916-24 (EudraCT Number)
Record Dates: First submitted 2011-08-03; First posted 2011-08-04 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Healthy Volunteer
MeSH Terms: interventions — Charcoal

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: RO4995819; Drug: activated charcoal
- 2 (Active Comparator)
  Interventions: Drug: RO4995819

INTERVENTIONS:
Drug: RO4995819 — single oral dose
Drug: activated charcoal — orally 3 times daily, Days 1-7
  Arms: 1

SUMMARY:
This open-label, two period crossover study will evaluate the effect of multiple doses of activated charcoal on the pharmacokinetics of a single oral dose of RO4995819 in healthy volunteers. Each enrolled subject will receive two single oral doses of RO4995819 separated by a wash-out period of up to 9 weeks. In period 1, subjects will receive concomitantly with the single dose of RO4995819 multiple oral doses of activated charcoal until Day 7. In period 2, only a single dose of RO4995819 but no activated charcoal will be administered.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects, 18 to 65 years of age, inclusive
* Body mass index (BMI) 18 to 30 kg/m2 inclusive
* All subjects must agree to use a barrier method (e.g. condom) throughout the study and for up to 5 months after the last dose of study drug
* Significant past or present disorders of the central nervous system, psychiatric disorders or behavioral disturbances.

Exclusion Criteria:

* Any suspicion or history of alcohol abuse and/or consumption of other drugs of abuse
* Positive for hepatitis B, hepatitis C, or HIV 1 or HIV 2
* Participation in an investigational drug or device study within 3 months prior to first administration of the study drug
* Any confirmed allergic reaction against any drug or multiple allergies
* Dietary restrictions that would prohibit the consumption of standardized meals
* Positive cotinine test and/or any use of nicotine containing products
* Clinically relevant history of constipation or bowel disorder
* Known intolerability to activated charcoal

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2011-08; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
C max: maximum observed plasma concentration | 18 weeks
T max: time of maximum observed plasma concentration | 18 weeks
T1/2: apparent terminal half-life | 18 weeks
AUC: area under the plasma concentration-time curve | 18 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- Rennes, France